CLINICAL TRIAL: NCT06390969
Title: A Survey on the Practice and Interpretation of Various Diagnostic Tests for Tuberculous Pleuritis Among Respiratory Physicians
Brief Title: TBP Survey Among Respiratory Physicians
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: TBP_survey
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Pleural Effusion; Tuberculosis, Pleural
MeSH Terms: conditions — Pleural Effusion; Tuberculosis, Pleural | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey respondent: All respiratory doctors who respond to the survey
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Cross-sectional online survey

SUMMARY:
Tuberculosis is a major infectious disease with a high mortality burden in the Asia-Pacific region and worldwide. Among various types of extrapulmonary tuberculosis, tuberculous pleuritis (TBP) is amongst the most common manifestations. TBP is also a major underlying cause among patients hospitalised with new-onset unilateral pleural effusion. The workup of TBP frequently involves thoracentesis to retrieve pleural fluid and pleural biopsy for microbiological and histological interpretations. However, the diagnostic accuracy of these tests is of unsatisfactory sensitivity, making diagnosing TBP challenging. In addition, certain tests, including pleural fluid adenosine deaminase (ADA), Mycobacterium tuberculosis polymerase chain reaction (MTB PCR), advanced biopsy procedures (e.g. real-time image-guided biopsy, pleuroscopy) are not readily available in developing regions due to scarcity of resources and lack of expertise. All these factors lead to heterogeneous practice in approaching new-onset pleural effusion, interpretation of pleural TB investigations, and timing of TBP treatment initiation among respiratory physicians in different Asia-Pacific regions. The proposed multinational survey aims to understand the real-world clinical practice in approaching patients with new-onset unilateral pleural effusion and diagnosing TBP in Asia-Pacific regions with intermediate to high TB burden. The results will reflect the current practice of diagnosing TBP, clinical and resource discrepancies in investigating TBP, management of TBP and help prioritise the need for further research in TBP

DETAILED DESCRIPTION:
Tuberculosis (TB) is one of the major global health threats, with an estimated 10.6 million people infected with TB in 2021, with 1.6 million dying from the disease. Apart from pulmonary involvement as the major manifestation of TB, there is an increasing trend of extrapulmonary TB (EPTB) reported in different continents. Among EPTB, TB pleuritis (TBP) was the most prevalent form in several large Chinese retrospective studies.

Diagnosing TBP is challenging due to paucibacillary involvement (TB disease caused by a small number of bacteria) of the pleural space. A diagnosis of definite TBP can be secured if the acid-fast bacilli (AFB), Mycobacterium tuberculosis (MTB) culture of pleural fluid reveals positive results. However, these conventional diagnostic tests for TBP are insufficiently sensitive, and the long turnaround time of culture would also delay the initial clinical management. The diagnosis of definite TBP may also be based on compatible histological findings of the pleural tissue obtained by biopsy procedures (bedside biopsy by Abram's needle, real-time image-guided biopsy by radiologists or experienced respiratory physicians, or pleuroscopy). The availability and waiting time of these procedures vary in different regions. Due to these reasons, a diagnosis of probable TBP may be pursued instead. This diagnostic entity is based on compatible clinical presentations with exudative, lymphocytic pleural effusion and raised pleural fluid biomarkers, commonly adenosine deaminase (ADA), without diagnostic microbiological results and alternative clinical explanation [10]. Other than pleural fluid ADA, several pleural fluid biomarkers have been explored to assist in diagnosing probable TBP. Therefore, a significant proportion of patients suspected to have TBP may have empirical anti-TB treatment initiated in the absence of a confirmatory diagnosis. In addition, these diagnostic clinical challenges are magnified among Asia-Pacific developing countries where contemporary diagnostic tools may be unavailable and hinder local TB control.

There is a lack of regional Asia-Pacific real-world evidence of how TBP is diagnosed and how pleural fluid biomarkers are used. We hypothesise that heterogeneous practice towards new-onset unilateral pleural effusion and understanding different diagnostic tests for diagnosing TBP across different countries depends on the TB burden and availability of advanced pleural services. Therefore, a multinational survey study is designed to understand the real-world practice of managing new-onset unilateral pleural effusion, the availability and utilisation of different diagnostic tests for TBP, and the factors determining the timing of initiating empirical anti-TB treatment for TBP among respiratory physicians in the Asia-Pacific region.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory doctors practising in Asia-Pacific region

Exclusion Criteria:

* Do not consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The questionnaire will be sent via social media, including WhatsApp, Facebook, X (formerly known as Twitter), targeting respiratory physicians practising in various Asia-Pacific regions, especially regions with intermediate to high TB burden, through snowball sampling. These regions include China, Hong Kong, India, Malaysia, Philippines, Singapore, Taiwan (based on the network of the applicants) and beyond.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Treatment decision | 1 month
  the proprtion of respondents that would consider TBP as one of the differential diagnoses when approaching new-onset unilateral pleural effusion

SECONDARY OUTCOMES:
Test availability | 1 month
  To evaluate the availability of different diagnostic tests for diagnosing TBP, in 5 point Likert scale
Disease understanding | 1 month
  To evaluate the understanding and utilisation of pleural fluid biomarkers for TBP among respiratory physicians, in 5 point Likert scale
Treatment decision for suspected tuberculosis | 1 month
  To evaluate the factors determining the initiation of empirical anti-TB treatment for probable TBP, in 5 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Director — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No